CLINICAL TRIAL: NCT06728072
Title: Pilot Study Evaluating Microbiome Modulation Therapy (MBMT) With Ciprofloxacin, Metronidazole, and Aspirin in Addition to Standard of Care Chemotherapy in Patients Undergoing First-Line Therapy for Metastatic Colorectal Cancer
Brief Title: Addition of Antibiotics to Upfront Treatment Regimen for Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-23-20875; HM20031481 (Other: Virginia Commonwealth University)
Record Dates: First submitted 2024-11-07; First posted 2024-12-11 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Colorectal Cancer; CRC
Keywords: Colorectal Cancer; CRC
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Metronidazole; Ciprofloxacin; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard of care (No Intervention): First line chemotherapy as directed. Standard of care chemotherapy treatment options include but are not limited to the following:
  * FOLFOX every 2 weeks
  * FOLFIRI every 2 weeks
  * FOLFOX + bevacizumab or panitumumab every 2 weeks
  * FOLFIRI + bevacizumab or panitumumab every 2 weeks
  * CAPEOX every 3 weeks
  * CAPEOX + bevacizumab or panitumumab every 3 weeks
- Metronidazole Ciprofloxacin and Aspirin Therapy (Experimental): First line chemo therapy (standard of care) + Microbiome modulation therapy MBMT 500 mg metronidazole 3 times daily, 500 mg ciprofloxacin twice daily, and 81 mg aspirin once daily for 28 days
  Interventions: Drug: Standard of Care Chemotherapy + Metronidazole, ciprofloxacin, aspirin

INTERVENTIONS:
Drug: Standard of Care Chemotherapy + Metronidazole, ciprofloxacin, aspirin — Metronidazole, ciprofloxacin, aspirin is initiated Cycle 1 Day 1 of chemotherapy. May be initiated any time from 7 days before Cycle 1 Day 1 up to and including Cycle 1 Day 3
  Arms: Metronidazole Ciprofloxacin and Aspirin Therapy

SUMMARY:
This is a 2-arm, noncomparative phase 2 trial designed to evaluate treatment outcomes with or without the addition of ciprofloxacin, metronidazole, and aspirin to first-line chemotherapy for patients with stage IV colorectal cancer (CRC).

DETAILED DESCRIPTION:
This is a pilot study to evaluate the efficacy and safety of chemotherapy with or without MBMT in patients with metastatic CRC. The primary objective is to evaluate the efficacy, as determined by the ORR, of fluorouracil (5FU) based treatment regimen with and without MBMT in patients with CRC.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage IV colorectal cancer
* Measurable disease by Response evaluation criteria in solid tumors (RECIST) 1.1 criteria
* Planned first-line treatment with a 5FU-based doublet chemotherapy regimen for colon cancer, specifics of the regimen at the discretion of the treating physician Note: Patients who have received adjuvant therapy >6 months prior are eligible
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2
* Absolute neutrophil count (ANC) ≥1,500 cells/μL
* Platelet count ≥100,000 cells/μL
* Hemoglobin ≥8 g/dL Note: The use of transfusion or other intervention to achieve hemoglobin ≥8 g/dL is acceptable.
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 × upper limit of normal (ULN) Note: Patients with documented liver metastases: AST and ALT ≤5 × ULN
* Serum creatinine ≤1.5 x ULN or calculated creatinine clearance ≥40 mL/min using the Cockcroft-Gault equation: (140 - age) × body weight/plasma creatinine × 72 (× 0.85 if female)
* Radiographically measurable disease by RECIST 1.1
* Nonpregnant and not actively breastfeeding
* Sexually active patients of childbearing potential and their partners must agree to use medically acceptable form of contraception, per treating investigator, throughout the study Patients should continue to use medically acceptable methods of contraception after study treatment ends, following the guidance for their specific chemotherapy regimen.

Childbearing potential excludes:

Age > 50 years and naturally amenorrhoeic for > 1 year OR previous hysterectomy or bilateral salpingo-oophorectomy

* Patients on a pre-existing daily aspirin regimen may participate in the study without interrupting this regimen.
* Patients with a contraindication to aspirin may participate in the study. These patients will not be required to take aspirin as part of the study treatment.

Exclusion Criteria:

* Total colectomy
* Diagnosed with Cockayne Syndrome
* Using disulfiram, tizanidine, or theophylline and unable to stop taking these medications for the length of the microbiome modulation therapy
* On methotrexate doses of 15 mg/week or more
* History of allergic reaction to ciprofloxacin, metronidazole, or aspirin
* Fuss course of antibiotics in the 30 days before chemotherapy start Note: Full course is defined as ≥5 doses with an intent to treat a defined infection. Use of antibiotics intended for prophylaxis at the time of surgery is allowed
* Corrected QT interval (QTc) >480 on baseline ECG
* Diagnosed with a malabsorptive syndrome
* Inability to swallow tablets

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2035-07-01 (Estimated); Study Completion 2035-07-01 (Estimated)

PRIMARY OUTCOMES:
Best response by analysis using Response Evaluation Criteria in Solid Tumors | Up to 5 years
  Evaluate the objective response rate (ORR) of a fluorouracil (based) treatment regimen with or without the addition of MBMT in patients with colorectal cancer (CRC) by the number of participants that have a partial (PR) or complete response (CR) using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) criteria.

SECONDARY OUTCOMES:
Estimate the overall survival (OS) of patients with colorectal cancer (CRC) treated with a 5FU-based treatment regimen with or without the addition of MBMT. | Up to 5 years
  Evaluate the overall participant survival (OS) defined as the duration of time from diagnosis to date of death by any cause.
Estimate the progression free survival (PFS) of patients with CRC treated with a 5FU-based treatment regimen with or without the addition of the MBMT | Up to 5 years
  Progression free survival (PFS) is defined as the duration of time from start of study 5FU-based treatment regimen to date of first progression or relapse.
Assess the tolerability of the study antibiotic regimen | Day 28 +/- 7 days
  Total number of antibiotic doses over 28 days
Assess the tolerability of the study aspirin regimen for the duration of chemotherapy | Day 28 +/- 7 days
  Total number of aspirin doses over 28 days
Evaluate the safety of MBMT in addition to a 5FU-based treatment regimen | Beginning of study procedures through day 28 Non-interventional arm), through day 90 (interventional arm)
  The number of Adverse Events (AEs) captured using criteria in the National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE v5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Kinsey, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No